CLINICAL TRIAL: NCT03542240
Title: Effects of Curcumin Supplementation on Gut Barrier Function in Patients With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HM20012060
Record Dates: First submitted 2018-05-18; First posted 2018-05-31 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Obesity; High Blood Pressure; High Cholesterol; Type2 Diabetes; Heart Diseases
Keywords: curcumin; microbiome; dietary supplements; gut bacteria
MeSH Terms: conditions — Obesity; Hypertension; Hypercholesterolemia; Heart Diseases | interventions — Curcumin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Curcumin (Experimental)
  Interventions: Dietary Supplement: Curcumin

INTERVENTIONS:
Dietary Supplement: Curcumin — 500 milligram daily supplement

SUMMARY:
This study will investigate the effects of curcumin on the structure/function of the body by investigating whether targeted improvement of intestinal barrier function by supplementation with oral curcumin will result in attenuation of lipopolysaccharide (LPS) translocation and/or intestinal inflammation.

DETAILED DESCRIPTION:
A typical diet in the United States, also known as Western diet, is very high in sugars and saturated fat, and poor in food such as fruits, vegetables, fish and whole grains. This type of diet is associated with higher risk to develop obesity and other health problems such as high blood pressure, high cholesterol, Type 2 diabetes, and heart disease. Western diet can also cause changes in the gut that allow bacteria that are typically only present in the gut to leak out into the bloodstream. It is thought that having gut bacteria in the bloodstream may play a role in the development of diseases like Type 2 diabetes and heart disease.

Curcumin is a dietary supplement that comes from the root of the turmeric plant, and it may have an effect on the function of the gut and the leakage of gut bacteria into the bloodstream. The purpose of this research study is to evaluate the effects of daily curcumin dietary supplements on the function of the gut in subjects who are at risk for cardiovascular and metabolic diseases, for example they have increased blood pressure, increase waist circumference and high triglycerides (fat in the blood).

ELIGIBILITY:
Inclusion Criteria:

1. Based on National Institutes of Health (NIH) definition of Metabolic syndrome, the subject must meet at least 3 of the following criteria:

   A. Waist Circumference: Female ≥ 88 cm, Male ≥ 102 cm B. Blood Pressure: ≥ 130/85 mm/Hg and/or treatment with blood pressure lowering medication C. Impaired fasting glucose or HbA1c (fasting glucose ≥ 100 mg/dl or HgA1c ≥ 5.7 D. HDL-C: Females< 50 mg/dl, Males < 40 mg/dl E. Triglycerides ≥ 150 mg/dl
2. Willing and able to comply with the study protocol

Exclusion Criteria:

1. Diabetes
2. Established cardiovascular disease
3. Pre-existing liver disease other than NAFLD
4. Chronic kidney disease (Stage 4 and 5)
5. Rheumatological disease
6. Active malignancy
7. Alcohol consumption greater than 7 drinks per week for females and greater than 14 drinks per week for males
8. Current use of metformin and/or steroids
9. Curcumin supplementation
10. Females of child-bearing potential (NOT of child-bearing potential is defined as s/p hysterectomy or post-menopausal.)
11. Prisoners/wards of the state and individuals with limited English proficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2020-11-13 (Actual)

PRIMARY OUTCOMES:
Change inintestinal permeability | Baseline to 12 months
  Measured by level plasma lipopolysaccharide (LPS). A reduction in LPS suggests a reduction in intestinal permeability
Change in intestinal barrier function | Baseline to 12 months
  Measured by level of excreted Zonulin in stool samples. A reduction in Zonulin suggests a reduction in intestinal barrier function

CONTACTS AND LOCATIONS:
Overall Officials: Susan Wolver, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States